CLINICAL TRIAL: NCT06448455
Title: Observation of Frailty in Lung Cancer Patients and Its Influencing Factors
Brief Title: Observation on the Frailty Status of Lung Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Wang Jing, Head nurse, Peking University Third Hospital
Other Study IDs: LM2024248
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Frailty; Factor
MeSH Terms: conditions — Lung Neoplasms; Frailty | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung cancer patients: Through convenience sampling, lung cancer patients who were hospitalized and outpatients in the cancer chemotherapy Department of Peking University Third Hospital were selected as the research objects of this study.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Collect relevant data of patients

SUMMARY:
Using the Integrated Conceptual Model of Frailty (ICMF) and Frailty Framework among Vulnerable Population (FFVP) as theoretical basis, the frailty status of lung cancer patients is described, and the physiological, psychological, and social frailty of lung cancer patients are comprehensively evaluated and analyzed. The influencing factors related to frailty are explored, in order to provide a basis for effective intervention research on lung cancer patients in the future.

DETAILED DESCRIPTION:
The frailty of lung cancer patients is the result of multiple systems and factors, and its pathological and physiological changes include neuroendocrine disorders, malnutrition, sarcopenia, chronic inflammatory reactions, etc., accompanied by comorbidities and aging, and various factors promote the occurrence of frailty. Previous studies have found that older age, female gender, low education level, multiple drug use, smoking, lack of exercise, comorbidities, falls, sleep disorders, and anxiety and depression are the influencing factors of frailty in the elderly . When many domestic scholars study the frailty characteristics of elderly lung cancer patients, they have found that patients with advanced age, low BMI, divorce or widowhood, smoking, higher lung cancer staging, comorbidities with other diseases, multiple medications, poor nutrition, lower daily living ability, long disease course, depression, and lower red blood cells, albumin, and hemoglobin are more prone to frailty .

In summary, lung cancer patients are at risk of frailty, with a high incidence and an impact on the occurrence of adverse health outcomes. The conclusions drawn from different studies regarding the incidence and measurement of frailty in lung cancer patients vary. The frailty of lung cancer patients is influenced by multiple factors, not only involving demographic and disease-related factors. At present, there is limited research both domestically and internationally, mainly focusing on the impact of frailty in lung cancer patients on adverse health outcomes. There is a lack of research on the current situation and related factors of frailty in lung cancer patients. Most studies have explored demographic and disease-related factors in lung cancer patients, with little involvement in other variables such as psychological and social factors. Given the significant importance of frailty intervention in improving the health status of lung cancer patients, it is necessary to comprehensively evaluate the frailty status and related factors of lung cancer patients. Therefore, this study intends to use the Integrated Conceptual Model of Frailty (ICMF) and Frailty Framework among Vulnerable Population (FFVP) as theoretical basis to describe the frailty status of lung cancer patients, comprehensively evaluate and analyze the physiological, psychological, and social frailty of lung cancer patients, and explore the influencing factors related to frailty, in order to provide a basis for effective intervention research on lung cancer patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Lung cancer was diagnosed by pathology or cytology;
* Age ≥ 18 years;
* Be able to complete this questionnaire independently or under the guidance of the researcher;
* Informed consent and voluntary participation in this study.

Exclusion Criteria:

* Serious physical diseases (heart, lung, kidney and other important organ failure);
* Patients with a history of dementia, mental illness, intellectual disability, and cognitive impairment;
* Blind, deaf and aphasic patients;
* Participate in other studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will select lung cancer patients who are hospitalized and outpatients in the cancer chemotherapy Department of Peking University Third Hospital as the research object through convenient sampling.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Frailty | First day of admission
  Filburg Frailty Indicator，The score range is 0-55 points, and patients with ≥ 2points are diagnosed as debilitated. The higher the score of the total scale, the more serious the weakness.

SECONDARY OUTCOMES:
Sleep Quality | First day of admission
  Pittsburgh Sleep Quality Index，The total score in the table ranges from 0 to 21 points. The higher the score, the worse the sleep quality.
Anxiety | First day of admission
  Hospital Anxiety Scales，The scores range from 0 to 21. The higher the score, the more serious the anxiety.
Depression | First day of admission
  Hospital Depression Scales，The scores range from 0 to 21. The higher the score, the more serious the depression.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wang, Principal Investigator — Peking University Third Hospital Library
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available on reasonable request from the corresponding author. The data are not publicly available due to privacy or ethical restrictions.

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Shi JF, Wang L, Wu N, Li JL, Hui ZG, Liu SM, Yang BY, Gao SG, Ren JS, Huang HY, Zhu J, Liu CC, Fan JH, Zhao SJ, Xing PY, Zhang Y, Li N, Lei WD, Wang DB, Huang YC, Liao XZ, Xing XJ, Du LB, Yang L, Liu YQ, Zhang YZ, Zhang K, Qiao YL, He J, Dai M; LuCCRES Group. Clinical characteristics and medical service utilization of lung cancer in China, 2005-2014: Overall design and results from a multicenter retrospective epidemiologic survey. Lung Cancer. 2019 Feb;128:91-100. doi: 10.1016/j.lungcan.2018.11.031. Epub 2018 Nov 24. PMID 30642458
- [Result] Ruiz J, Miller AA, Tooze JA, Crane S, Petty WJ, Gajra A, Klepin HD. Frailty assessment predicts toxicity during first cycle chemotherapy for advanced lung cancer regardless of chronologic age. J Geriatr Oncol. 2019 Jan;10(1):48-54. doi: 10.1016/j.jgo.2018.06.007. Epub 2018 Jul 10. PMID 30005982
- [Result] Komici K, Bencivenga L, Navani N, D'Agnano V, Guerra G, Bianco A, Rengo G, Perrotta F. Frailty in Patients With Lung Cancer: A Systematic Review and Meta-Analysis. Chest. 2022 Aug;162(2):485-497. doi: 10.1016/j.chest.2022.02.027. Epub 2022 Feb 22. PMID 35217002
- [Result] Duan L, Cui H, Zhang W, Wu S. Symptoms and experiences of frailty in lung cancer patients with chemotherapy: A mixed-method approach. Front Oncol. 2022 Oct 6;12:1019006. doi: 10.3389/fonc.2022.1019006. eCollection 2022. PMID 36276107